CLINICAL TRIAL: NCT04526301
Title: Home With TablO outcoMEs (HOME) Registry
Acronym: HOME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Outset Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-02
Record Dates: First submitted 2020-08-14; First posted 2020-08-25 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-08

CONDITIONS: End Stage Renal Disease
Keywords: Tablo; Outset Medical; ESRD; Home Hemodialysis; HHD; ESKD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Tablo Hemodialysis System: Home dialysis treatment with the Tablo Hemodialysis System
  Interventions: Device: Tablo Hemodialysis System

INTERVENTIONS:
Device: Tablo Hemodialysis System — Home hemodialysis treatments ~4 times a week.

SUMMARY:
Prospective, multicenter, single arm, post-market study to evaluate real world clinical outcomes in ESRD patients receiving in-home dialysis on the Tablo Hemodialysis System.

ELIGIBILITY:
Inclusion Criteria:

* Participant (patient and/or care partner) is at least 15 years of age and has provided informed consent and has signed a Health Insurance Portability and Accountability Act of 1996 (HIPAA) compliant authorization statement.
* Participant weighs ≥ 34kg.
* Participant has end stage renal disease (ESRD) adequately treated by maintenance dialysis.
* Participant plans to start or has started home treatment (≤ 6 months) with the Tablo Hemodialysis System.
* Participant is willing and able to comply with the Protocol requirements and perform all site required treatments and clinical evaluations.

Exclusion Criteria:

* Participant and/or care partner is unable to read English or Spanish.
* Participant has a home environment that is deemed inappropriate for home dialysis.
* Participant and/or care partner is unable to successfully complete the Tablo training program
* Participant is pregnant or plans to become pregnant.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with end stage renal disease (ESRD) who are on, or planning to be on, maintenance hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-14 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Weekly Standardized Dialysis Adequacy | 12-months
  Weekly standardized dialysis adequacy (stdKt/V) measured using the second-generation formula of Daugirdas. This formula normalizes urea clearance among heterogeneous hemodialysis schedules, where K=dialyzer clearance or urea, t=treatment time, and V=subject's volume of urea distribution. stdKt/V values of ≥ 2.1 are regarded as being adequate.

OTHER OUTCOMES:
Health Outcomes | Change from Baseline at 12-months
  Change in health outcomes from baseline to 12-months, as measured by the 12-item Short Form Health Survey (SF-12) Questionnaire. The questionnaire consists of 12 items weighted and summed to provide physical and mental health scores (PCS and MCS). The two composite scores are computed using the scores on twelve questions that range from 0 to 100. Higher scores mean a better outcome.
Sleep Outcomes | Change from Baseline at 12-months
  Change in sleep from baseline to 12-months, as measured by the Insomnia Severity Index (ISI). The minimum and maximum values are 0 and 28 scores, respectively. Higher scores mean a worse outcome.
Care Partner Burden | Change from Baseline at 12-months
  Change in care partner burden from baseline to 12-months, as measured by the Zarit Burden Interview-12 (ZBI-12) scale. The scale score is calculated by summing each item to produce a total score between 0 and 24, with higher scores indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Satellite Healthcare, Inc., San Jose, California
  - Desert Cities Dialysis, Victorville, California
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - St. Peter's Health, Helena, Montana
  - Dialysis Center of Lincoln, Lincoln, Nebraska
  - Parker Jewish Institute, New Hyde Park, New York
  - NYU Grossman School of Medicine, New York, New York
  - Rogosin Institute, New York, New York
  - USRC Kidney Research, Plano, Texas
  - University of Virginia, Staunton, Virginia

IPD SHARING:
Plan to Share IPD: No